CLINICAL TRIAL: NCT05243706
Title: Evaluation of The Effect of Loratadine Versus Diosmin/Hesperidin Combination on Vinca Alkaloids Induced Neuropathy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Noha Kamal Morsy Ibraheem, Assistant lecturer at faculty of Pharmacy, University of Sadat City, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AinShamsU2
Record Dates: First submitted 2022-01-22; First posted 2022-02-17 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Vinca Alkaloid Adverse Reaction
Keywords: neuropathy; Vinca alkaloids; Diosmin/Hespridin; Loratadine
MeSH Terms: interventions — Loratadine; Diosmin; Hesperidin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group (No Intervention): 30 patients will receive Vincristine 1.5 mg/m2 (maximum: 2 mg) or Vinblastine 6 mg/m2 according to treatment protocol.
- Loratadine group (Experimental): 30 patients will receive One tablet 10 mg orally once daily starting with vincristine or vinblastine administration for three cycles
  Interventions: Drug: Loratadine
- diosmin 450mg / hesperidin 50 mg group (Experimental): 30 patients will receive 50 mg Hesperidin and Micronized purified flavonoid fraction (MPFF) 450 diosmin combination one film coated tablet orally twice daily starting with vincristine or vinblastine administration for three cycles
  Interventions: Drug: Diosmin/ Hesperidin

INTERVENTIONS:
Drug: Loratadine — Intervention is given to study its' effect on vinca alkaloids induced neuropathy
  Arms: Loratadine group
Drug: Diosmin/ Hesperidin — Intervention is given to study its effect on vinca alkaloids induced neuropathy
  Arms: diosmin 450mg / hesperidin 50 mg group

SUMMARY:
All vinca alkaloids causes neuropathy. The incidence of peripheral neuropathy is 30 %-40 % in patients treated with vincristine. The incidence of long term neurological adverse events from vinblastine ranged from 50% to 97%. In this study, the investigators will study the effect of using either loratadine or diosmin 450mg/ hesperidin 50 mg combination on neuropathy caused by Vinca alkaloids therapy. This study is a prospective, controlled, randomized, interventional and open-label clinical trial.

DETAILED DESCRIPTION:
Ninety patients will be randomly assigned to three groups as follows:

Group 1 (Control group): 30 patients will receive Vincristine 1.5 mg/m2 (maximum: 2 mg) or Vinblastine 6 mg/m2 according to treatment protocol.

Group 2 (Loratadine group): 30 patients will receive One tablet 10 mg orally once daily starting with vincristine or vinblastine administration for three cycles.

Group 3 (hesperidin 50 mg/diosmin 450mg group): 30 patients will receive 50 mg Hesperidin and Micronized purified flavonoid fraction (MPFF) 450 diosmin combination one film coated tablet orally twice daily starting with vincristine or vinblastine administration for three cycles .

Vincristine or Vinblastine dose will be adjusted as follows: Serum bilirubin 1.5 to 3 mg/dL or transaminases 2 to 3 times ULN or alkaline phosphatase increased: Administer 50% of dose.

Treatment allocation will follow a predefined randomization list and it will be computer generated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients prescribed vincristine or vinblastine according to standard protocols.
2. Adult patients older than18 years.
3. Patients willing to participate in the study and sign the informed consent.
4. Adequate bone barrow function (platelet count> 150 *103per microliter, absolute neutrophil count> 500 per microliter)
5. Eastern cooperative oncology group (ECOG) performance status Grade 0-2

Exclusion Criteria:

1. Hypersensitivity or contraindication to loratadine, hesperidin or diosmin combination or any component of the formulation.
2. Pre-existence or history of peripheral neuropathy due to a cause different from Vinca alkaloids induced neuropathy.
3. Receiving any other medication known to cause neuropathy.
4. Receiving medications with drug interaction grade X with Loratadine as Thalidomide, Tiotropium or Orphenadrine.
5. Women of childbearing potential not using an effective contraceptive method.
6. Pregnancy or breastfeeding.
7. Inability to understand patients' information and informed consent form.
8. Severe hepatic impairment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Assessing the efficacy of loratadine or diosmin 450mg/ hesperidin 50 mg on neuropathy pain intensity of Vinca alkaloids neuropathy compared to routine practice. | At baseline and after three cycles of vinca alkaloids (each cycle is 28 days)
  Measure of average pain intensity assessed by Numeric Pain Rating Scale (NS) change from baseline to after three cycles of vinca alkaloids therapy
Assessing the efficacy of loratadine or diosmin 450mg/ hesperidin 50 mg on pain quality (i.e. sensory and pain) of Vinca alkaloids neuropathy compared to routine practice. | At baseline and after three cycles of vinca alkaloids (each cycle is 28 days)
  Neuropathic Pain in 4 questions (DN4) change from baseline to after three cycles of vinca alkaloids therapy
Assessing the efficacy of loratadine or diosmin 450mg/ hesperidin 50 mg on symptoms of peripheral neuropathy of Vinca alkaloids compared to routine practice. | At baseline and after three cycles of vinca alkaloids (each cycle is 28 days)
  Functional Assessment of Cancer Therapy/Gynecologic Oncology Group - Neurotoxicity (FACT/GOG-NTX) change from baseline to after three cycles of vinca alkaloids therapy
Assessing the efficacy of loratadine or diosmin 450mg/ hesperidin 50 mg on development of Vinca alkaloids neuropathy compared to routine practice. | At baseline and after three cycles of vinca alkaloids (each cycle is 28 days)
  Measuring Peripheral blood Neurofilament Proteins and IL-1 beta change from baseline to after three cycles of vinca alkaloids therapy

SECONDARY OUTCOMES:
Evaluating the effect of loratadine versus diosmin 450mg/hesperidin 50 mg on the time to onset of neuropathy caused by Vinca alkaloids compared to control group. | from baseline to after Three cycles of vinca alkaloids (each cycle is 28 days)
  Measure the time of neuropathy onset in patients
Evaluating the Number of participants with Adverse Events of loratadine versus hesperidin 50 mg/diosmin 450mg by monitoring patients for undesirable effects | from baseline to after Three cycles of vinca alkaloids (each cycle is 28 days)
  The number of patients developing neuropathy as defined by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE)

IPD SHARING:
Plan to Share IPD: No